CLINICAL TRIAL: NCT06122103
Title: Comparison of Visual Outcomes With Mini-Monovision Between a Monofocal and an Adjustable Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Gainesville Eye Associates (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: CB-23-02
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Clareon Monofocal
  Interventions: Device: Clareon Monofocal
- Light-Adjustable Lens
  Interventions: Device: Light-Adjustable Lens

INTERVENTIONS:
Device: Clareon Monofocal — Clareon Monofocal Intraocular Lens (toric and non-toric)
  Groups: Clareon Monofocal
Device: Light-Adjustable Lens — Light-Adjustable Lens (Intraocular Lens)
  Groups: Light-Adjustable Lens

SUMMARY:
This study is a single center, multi-surgeon, prospective, randomized, comparative study of binocular corrected distance visual acuity (CDVA) after successful bilateral cataract surgery. Subjects will be assessed pre-operatively, operatively and at up to 6 postoperative visits. Clinical evaluations will include administration of patient reported spectacle usage questionnaire (PRSIQ), as well as measurement of monocular and binocular visual acuities at distance, intermediate, and near, defocus curve, manifest refraction, measurement of higher order aberrations.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet the following criteria: Note: Ocular criteria must be met in both eyes.

* Adult patients undergoing age-related cataract surgery with expected best- corrected visual outcomes of 20/25 or better
* Regular corneal astigmatism of 0.75D-2.50D
* Dilated pupil diameter of 7mm or greater

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Moderate-severe corneal pathology, irregular astigmatism, preexisting macular disease and other retinal degenerative diseases that is expected to cause future vision loss, glaucoma, severe dry eye disease, history of uveitis, ocular herpes simplex virus, nystagmus, strabismus, zonular laxity or dehiscence, pseudoexfoliation.
* History of corneal refractive and intraocular surgery.
* Patients taking systemic medication that may increase sensitivity to UV light or that may cause toxicity to the retina.

The principal investigator reserves the right to declare a patient ineligible or non- evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be adult normal astigmatic (≥ 0.75D corneal astigmatism) cataract patients presenting for cataract surgery who are considered appropriate candidates for intraocular lens implantation.
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton G Blehm, MD, Principal Investigator — Gainesville Eye Associates
Locations (1):
- Gainesville Eye Associates, Gainesville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Clareon Monofocal: Bilateral Implantation of the Clareon Monofocal IOL
- Light-Adjustable Lens: Bilateral Implantation of the Light-Adjustable Lens
Period: Overall Study
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Started | 70 | 68
Completed | 70 | 68
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clareon Monofocal | Light-Adjustable Lens | Total
Number analyzed (Participants) | 70 | 68 | 138
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.7 (7.9) | 70.8 (7.6) | 71.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 38 | 83
  Male | 25 | 30 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Binocular Corrected Distance Visual Acuity (CDVA)
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
logMAR | -0.03 (0.07) | -0.03 (0.07)

2. Secondary Outcome: Binocular Uncorrected Distance Visual Acuity (UDVA)
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
logMAR | 0.02 (0.09) | 0.03 (0.10)

3. Secondary Outcome: Binocular Distance Corrected Intermediate Visual Acuity (DCIVA)
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
logMAR | 0.17 (0.12) | 0.11 (0.11)

4. Secondary Outcome: Binocular Uncorrected Intermediate Visual Acuity (UIVA)
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
logMAR | 0.06 (0.11) | 0.04 (0.09)

5. Secondary Outcome: Monocular Corrected Distance Visual Acuity (CDVA)
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
Number analyzed (eyes) | 140 | 136
logMAR
  Dominant Eyes | -0.01 (0.07) | 0.01 (0.08)
  Non-Dominant Eyes | 0.02 (0.07) | 0.01 (0.07)

6. Secondary Outcome: Monocular Uncorrected Distance Visual Acuity (UDVA)
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
Number analyzed (eyes) | 140 | 136
logMAR
  Dominant Eyes | 0.05 (0.10) | 0.08 (0.12)
  Non-Dominant Eyes | 0.28 (0.18) | 0.26 (0.18)

7. Secondary Outcome: Monocular Distance Corrected Intermediate Visual Acuity (DCIVA)
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
Number analyzed (eyes) | 140 | 136
logMAR
  Dominant Eyes | 0.26 (0.12) | 0.23 (0.14)
  Non-Dominant Eyes | 0.25 (0.14) | 0.22 (0.13)

8. Secondary Outcome: Monocular Uncorrected Intermediate Visual Acuity (UIVA)
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
Number analyzed (eyes) | 140 | 136
logMAR
  Dominant Eyes | 0.30 (0.18) | 0.22 (0.16)
  Non-Dominant Eyes | 0.11 (0.13) | 0.08 (0.12)

9. Other Pre Specified Outcome: Binocular Distance-corrected Near Visual Acuity (DCNVA)
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
logMAR | 0.38 (0.17) | 0.34 (0.16)

10. Other Pre Specified Outcome: Binocular Uncorrected Near Visual Acuity (UNVA)
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
logMAR | 0.25 (0.16) | 0.18 (0.11)

11. Other Pre Specified Outcome: Monocular Distance Corrected Defocus Curve
Time Frame: 3 months postop
Population: Data were collected for Dominant and Non-Dominant Eyes for the LAL Group and Dominant Eyes for the Clareon Group
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
Number analyzed (eyes) | 140 | 136
logMAR
  1.00 D (Dominant Eyes): number analyzed (eyes) | 70 | 68
  1.00 D (Dominant Eyes) | 0.28 (0.16) | 0.24 (0.18)
  1.00 D (Non-Dominant Eyes): number analyzed (eyes) | 0 | 68
  1.00 D (Non-Dominant Eyes) |  | 0.30 (0.23)
  0.50 D (Dominant Eyes): number analyzed (eyes) | 70 | 68
  0.50 D (Dominant Eyes) | 0.12 (0.13) | 0.14 (0.20)
  0.50 D (Non-Dominant Eyes): number analyzed (eyes) | 0 | 68
  0.50 D (Non-Dominant Eyes) |  | 0.18 (0.22)
  0.25 D (Dominant Eyes): number analyzed (eyes) | 70 | 68
  0.25 D (Dominant Eyes) | 0.07 (0.12) | 0.10 (0.14)
  0.25 D (Non-Dominant Eyes): number analyzed (eyes) | 0 | 68
  0.25 D (Non-Dominant Eyes) |  | 0.14 (0.14)
  0.00 D (Dominant Eyes): number analyzed (eyes) | 70 | 68
  0.00 D (Dominant Eyes) | 0.03 (0.10) | 0.05 (0.12)
  0.00 D (Non-Dominant Eyes): number analyzed (Participants) | 0 | 68
  0.00 D (Non-Dominant Eyes): number analyzed (eyes) | 0 | 68
  0.00 D (Non-Dominant Eyes) |  | 0.10 (0.22)
  -0.25 D (Dominant Eyes): number analyzed (eyes) | 70 | 68
  -0.25 D (Dominant Eyes) | 0.07 (0.12) | 0.07 (0.10)
  -0.25 D (Non-Dominant Eyes): number analyzed (Participants) | 0 | 68
  -0.25 D (Non-Dominant Eyes): number analyzed (eyes) | 0 | 68
  -0.25 D (Non-Dominant Eyes) |  | 0.11 (0.20)
  -0.50 D (Dominant Eyes): number analyzed (eyes) | 70 | 68
  -0.50 D (Dominant Eyes) | 0.10 (0.12) | 0.10 (0.12)
  -0.50 D (Non-Dominant Eyes): number analyzed (eyes) | 0 | 68
  -0.50 D (Non-Dominant Eyes) |  | 0.13 (0.19)
  -1.00 D (Dominant Eyes): number analyzed (eyes) | 70 | 68
  -1.00 D (Dominant Eyes) | 0.21 (0.13) | 0.16 (0.14)
  -1.00 D (Non-Dominant Eyes): number analyzed (eyes) | 0 | 68
  -1.00 D (Non-Dominant Eyes) |  | 0.20 (0.16)
  -1.50 D (Dominant Eyes): number analyzed (eyes) | 70 | 68
  -1.50 D (Dominant Eyes) | 0.36 (0.16) | 0.30 (0.17)
  -1.50 D (Non-Dominant Eyes): number analyzed (eyes) | 0 | 68
  -1.50 D (Non-Dominant Eyes) |  | 0.28 (0.17)
  -2.00 D (Dominant Eyes): number analyzed (eyes) | 70 | 68
  -2.00 D (Dominant Eyes) | 0.48 (0.18) | 0.43 (0.19)
  -2.00 D (Non-Dominant Eyes): number analyzed (eyes) | 0 | 68
  -2.00 D (Non-Dominant Eyes) |  | 0.38 (0.19)
  -2.50 D (Dominant Eyes): number analyzed (eyes) | 70 | 68
  -2.50 D (Dominant Eyes) | 0.61 (0.19) | 0.58 (0.21)
  -2.50 D (Non-Dominant Eyes): number analyzed (eyes) | 0 | 68
  -2.50 D (Non-Dominant Eyes) |  | 0.50 (0.23)

12. Other Pre Specified Outcome: Binocular Distance Corrected Defocus Curve
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
logMAR
  1.00 D | 0.25 (0.14) | 0.22 (0.17)
  0.50 D | 0.08 (0.11) | 0.11 (0.12)
  0.25 D | 0.04 (0.09) | 0.07 (0.11)
  0.00 D | 0.00 (0.08) | 0.03 (0.09)
  -0.25 D | 0.03 (0.12) | 0.03 (0.09)
  -0.50 D | 0.05 (0.09) | 0.04 (0.09)
  -1.00 D | 0.09 (0.11) | 0.08 (0.12)
  -1.50 D | 0.11 (0.13) | 0.13 (0.13)
  -2.00 D | 0.13 (0.17) | 0.13 (0.15)
  -2.50 D | 0.21 (0.19) | 0.16 (0.21)

13. Other Pre Specified Outcome: Manifest Refraction
Description: MRSE, residual sphere, and residual astigmatism
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: D
Units Other Than Participants: eyes
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
Number analyzed (eyes) | 70 | 68
D
  Sphere (Dominant Eyes) | -0.13 (0.31) | -0.05 (0.24)
  Sphere (Non-Dominant Eyes) | -0.97 (0.29) | -1.08 (0.32)
  Cylinder (Dominant Eyes) | 0.06 (0.18) | 0.07 (0.19)
  Cylinder (Non-Dominant Eyes) | 0.06 (0.20) | 0.11 (0.22)
  MRSE (Dominant Eyes) | -0.10 (0.30) | -0.01 (0.24)
  MRSE (Non-Dominant Eyes) | -0.94 (0.31) | -1.03 (0.37)

14. Other Pre Specified Outcome: Patient Reported Spectacle Usage Questionnaire (PRSIQ)
Description: Participants are asked to indicate spectacle usage on a scale of "All of the time" to "None of the time" for distance, intermediate, and near vision.
Time Frame: 3 months postop
Population: Count of participants answering "None of the time" when asked "During the last 7 days, how often did you need glasses or contacts"
Measure: Number; unit: percentage of participants
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
percentage of participants
  Distance | 93 | 91
  Intermediate | 79 | 87
  Near | 37 | 49
  Overall | 39 | 50

15. Other Pre Specified Outcome: Wavefront Aberrometry Using iTrace (Internal, Ocular, and Corneal Total Higher Order Aberrations)
Description: Aberrometry was performed using the iTrace (Tracy Technologies, USA)
Time Frame: 3 months postop
Population: 70 dominant and 70 non-dominant eyes (140 eyes total) in the Clareon Group 68 dominant and 68 non-dominant eyes (136 eyes total) in the LAL Group
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: eyes
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
Number analyzed (Participants) | 70 | 68
Number analyzed (eyes) | 140 | 136
microns
  Ocular HOA (Dominant Eyes): number analyzed (eyes) | 70 | 68
  Ocular HOA (Dominant Eyes) | 0.36 (0.24) | 0.38 (0.21)
  Ocular HOA (Non-Dominant Eyes): number analyzed (eyes) | 70 | 68
  Ocular HOA (Non-Dominant Eyes) | 0.31 (0.23) | 0.45 (0.25)
  Internal HOA (Dominant Eyes): number analyzed (eyes) | 70 | 68
  Internal HOA (Dominant Eyes) | 0.25 (0.18) | 0.31 (0.16)
  Internal HOA (Non-Dominant Eyes): number analyzed (eyes) | 70 | 68
  Internal HOA (Non-Dominant Eyes) | 0.25 (0.26) | 0.40 (0.21)
  Corneal HOA (Dominant Eyes): number analyzed (eyes) | 70 | 68
  Corneal HOA (Dominant Eyes) | 0.29 (0.16) | 0.31 (0.20)
  Corneal HOA (Non-Dominant Eyes): number analyzed (eyes) | 70 | 68
  Corneal HOA (Non-Dominant Eyes) | 0.30 (0.22) | 0.37 (0.26)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Clareon Monofocal | Light-Adjustable Lens
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/68
Other Adverse Events (participants affected / at risk) | 6/70 | 14/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clareon Monofocal (N=70) | Light-Adjustable Lens (N=68)
YAG laser capsulotomy (Eye disorders) | 4 | 4
Dry Eye (Eye disorders) | 2 | 7
Herpes simplex virus keratitis (Eye disorders) | 0 | 2
Endophthalmitis (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT06122103/Prot_SAP_000.pdf